CLINICAL TRIAL: NCT01136395
Title: Impact of Rituximab Induction and Living Donation on Immunoregulation and Virus Control in Renal Transplantation - a Prospective Pilot Study
Brief Title: Impact of Rituximab (RTx) Induction and Living Donation on Immunoregulation and Virus Control in Renal Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Giessen (Other)
Collaborators: Heidelberg University (Other); German Cancer Research Center (Other); Astellas Pharma US, Inc. (Industry); Novartis (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Rolf Weimer, head of renal transplant program, University of Giessen, University of Giessen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NTx-RTx-LD-001; 2009-012198-36 (EudraCT Number)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Kidney Transplantation; Rituximab (RTx); Living Donors; Immunology; Virus
Keywords: Kidney Transplantation; Rituximab; Living Donor; ABO Incompatible (ABOi) Transplantation; Immunology; Cytomegalovirus (CMV); Epstein Barr virus (EBV); Polyomavirus
MeSH Terms: conditions — Virus Diseases; Epstein-Barr Virus Infections | interventions — Rituximab; Kidney Transplantation; Antibodies, Monoclonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LD kidney transplantation, ABOi (Active Comparator): Living donor (LD) kidney transplantation, ABO incompatible (ABOi); Immunosuppressive treatment: Tacrolimus (Tacr)/ Mycophenolate sodium (MPS), Basiliximab induction, Rtx induction
  Interventions: Drug: Rituximab; Procedure: living donor transplantation
- LD kidney transplantation, ABOc (Active Comparator): Living donor (LD) kidney transplantation, ABO compatible (ABOc); Immunosuppressive treatment: Tacr/MPS, Basiliximab induction
  Interventions: Procedure: living donor transplantation
- DD kidney transplantation (Active Comparator): Deceased donor (DD) kidney transplantation, ABO compatible; Immunosuppressive treatment: Tacr/MPS, Basiliximab induction
  Interventions: Procedure: deceased donor transplantation

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 4 weeks before ABOi LD transplantation
  Other Names: Blood group incompatible (ABOi) living donor (LD) renal transplantation; Anti-CD20 (cluster of differentiation 20) Monoclonal Antibody (MoAb)
  Arms: LD kidney transplantation, ABOi
Procedure: living donor transplantation — living donor transplantation (ABO compatible) to be compared with deceased donor transplantation (ABO compatible) in its impact on immunological parameters of graft outcome and on viral replication (CMV, EBV, BK/JC), respectively
  Other Names: Blood group compatible (ABOc) LD NTx
  Arms: LD kidney transplantation, ABOc; LD kidney transplantation, ABOi
Procedure: deceased donor transplantation — deceased donor transplantation (ABO compatible) to be compared with living donor transplantation (ABO compatible) in its impact on immunological parameters of graft outcome and on viral replication (CMV, EBV, BK virus (BKV), JC virus (JCV)), respectively
  Other Names: Deceased donor (DD) renal transplantation
  Arms: DD kidney transplantation

SUMMARY:
This project comprises immunological and virological analyses within a prospective clinical study of Rituximab (Rtx)-treated blood group incompatible living donor (LD) renal transplant recipients compared to blood group compatible LD recipients without Rtx induction, and of living donor compared to deceased donor renal transplant recipients treated with tacrolimus (Tacr)/mycophenolate sodium (MPS). Aim of this project is to assess short- and long-term effects of immunosuppressive therapy (Rtx induction) and of living donation on immunological and histological parameters of graft outcome and on viral replication (BK virus (BKV), JC virus (JCV), cytomegalovirus (CMV), Epstein Barr virus (EBV)) with the potential to improve long-term graft outcome and to enable risk estimation of virus disease.

DETAILED DESCRIPTION:
Objective. Blood group incompatible (ABOi) LD renal transplantation represents a recognized treatment modality in Germany. In this setting, ethical considerations allow for a detailed study of short- and long-term immunological and virological effects of Rtx induction therapy, including sequential protocol biopsies. In the proposed project we will perform analyses on peripheral blood, iliac lymph nodes and protocol biopsies. Protocol biopsies are routinely obtained 3 and 12 months posttransplant at the Universities of Giessen and Freiburg. In this prospective, open pilot study, immunological parameters of graft outcome and control of polyomavirus, EBV and CMV replication will be compared between RTx-treated ABOi LD renal transplant recipients (n=25-30, group 1) and blood group compatible LD renal transplant recipients without Rtx induction (n=25-30, group 2) but otherwise comparable immunosuppressive treatment (MPS and Tacr, switch to Tacr-MR (modified release) within 2 weeks posttransplant; follow-up of 5 years). The same analyses will be done in DD renal transplant recipients treated with Tacr (switch to Tacr-ME) and MPS (n=25-30, group 3). This study design allows to analyze the impact of living donation on immunoregulation and virus control (groups 2 versus 3).

Background. There is growing evidence that humoral mechanisms play a major role in chronic allograft dysfunction, which was shown to be significantly associated with de-novo formation of donor-specific antibodies against human leucocyte antigens (HLA). However, B cells appear to act not only in humoral responses against the graft but may play a significant role in T-cell mediated antidonor responses due to their role as effective antigen-presenting cells. This is further suggested by the fact that Rtx is effective in primarily T-cell mediated diseases such as rheumatoid arthritis or multiple sclerosis.

Hypothesis/specific aims. We hypothesize that Rtx induction may alter immunoregulation short- and long-term after renal transplantation with the potential to improve long-term outcome. Graft protective effects of Rtx induction may be provided by B cell depletion and the resulting effects on humoral as well as T cell responses, and also by altered responses after B cell repopulation. Possible negative effects of Rtx on polyomavirus and CMV control as well as protective effects on EBV replication, de-novo monoclonal gammopathy and regulation of lymphoma growth factors (interleukins 6 and 10 (IL-6, IL-10)) will be analyzed. Furthermore, B cell subset analysis in peripheral blood and the probably associated impact of Rtx on B cell depletion in graft draining iliac lymph nodes may enable us to establish an optimized Rtx dosage and thereby allow successful ABOi renal transplantation without the currently observed 15% drop outs.

Preliminary results. We have performed clinical studies showing the predictive power of immune parameters such as regulatory anti-Fab autoantibodies, sCD30, CD4 (cluster of differentiation 4) helper activity, and CD4 cell IL-4 (interleukin 4) and IL-10 (interleukin 10) responses on graft outcome. The long-term effect of Rtx induction therapy and of living donation on these parameters will be analyzed.

Previously, we found that patients at risk of polyomavirus nephropathy may be recognized early posttransplant by sequential reverse transcriptase polymerase chain (rt-PCR) assessment of polyomavirus replication in urine. Sequential rt-PCR testing of polyomavirus replication in urine and plasma will be used to analyze effects of Rtx induction on polyomavirus control.

Proposed methods. Immune parameters will be analyzed mainly pretransplant, 3 months and 1, 2 and 5 years posttransplant. Flow cytometry (including regulatory T cells, B cell subsets, expression of cytokine receptors, costimulatory and adhesion molecules), mitogen-stimulated allogeneic cocultures, protein-A plaque assay (B cell responses, CD4 helper activity), intracellular cytokine analysis of CD4+ and CD8+ (cluster of differentiation 8) T cells, B cells and monocytes, rt-PCR for virological studies (BKV, JCV, CMV, EBV) and immunofluorescent staining of iliac lymph nodes (obtained at time of transplantation) and protocol biopsies will be used. Donor-specific antibodies will be detected using lymphocytotoxicity, HLA class I and II ELISA and Luminex assays. Donor-specificity will be confirmed by T- and B-cell crossmatch with donor cells. Regulatory IgG (immunoglobulin G) and IgA (immunoglobulin A) anti-Fab autoantibodies, neopterin and sCD30 will be assessed by ELISA.

Expected results. We expect that Rtx induction will show an impact on immunological parameters of graft outcome, such as de-novo posttransplant antidonor HLA antibody formation. This pilot study may allow for improved long-term kidney graft outcome in recipients with immunologic risk parameters by virtue of patient-tailored immunosuppressive therapy. In ABOi renal transplantation, this study may prevent the current 15% drop out rates by allowing an optimized Rtx dosage based on the intended dose response analysis (B cell subset analysis in blood and graft draining lymph nodes). Furthermore, this study will allow risk estimation of Rtx administration with respect to CMV and polyomavirus replication, and may provide clues concerning protection against EBV replication and posttransplant lymphoproliferative disease. The latter point is of great clinical importance in patients with an enhanced PTLD (posttransplant lymphoproliferative disease) risk such as EBV negative recipients of EBV positive grafts.

ELIGIBILITY:
Inclusion Criteria:

* De-novo kidney transplantation
* Deceased donors (blood group compatible) and living donors (blood group incompatible / blood group compatible)
* First, second and third renal transplants
* Immunized and non-immunized graft recipients
* Age of recipients 18 years or older
* Negative pregnancy test before transplantation

Exclusion Criteria:

* Contra-indications to use Tacr and MPS, respectively
* Contra-indications to use Rtx in the group of ABOi LD transplants
* Chronic hepatitis B, C or HIV infection
* Recurrent infectious disease
* Previous hepatitis B, if no prophylactic antiviral therapy is used
* Previous tuberculosis
* Hemoglobin<8,5g/dl, thrombocytes<80.000/ul or leucocytes<3000/ul
* Previous vaccination with a living vaccine <4 weeks pretransplant
* Significant enterogastric disease such as diverticulitis (contra-indicates MPS treatment)
* Children and adolescents (age less than 18 years)
* Pregnancy and breast-feeding women
* Refusal of an effective contraception in women capable of bearing children
* Combined transplantations such as simultaneous islet/kidney transplants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Impact of Rtx on immune parameters predictive of graft outcome including B cell responses | 5 years posttransplant
  immune parameters of graft outcome: see "detailed description"
Impact of living donation on immune parameters predictive of graft outcome including B cell responses | 5 years posttransplant
  parameters of graft outcome: see "detailed description"
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: EBV PCR (in blood)
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: CMV PCR (in blood)
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: BKV PCR (in blood)
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: BKV PCR (in urine)
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: JCV PCR (in blood)
Impact of Rtx on virus replication | 5 years posttransplant
  outcome measure description: JCV PCR (in urine)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: EBV PCR (in blood)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: CMV PCR (in blood)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: BKV PCR (in blood)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: BKV PCR (in urine)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: JCV PCR (in blood)
Impact of living donation on virus replication | 5 years posttransplant
  outcome measure description: JCV PCR (in urine)

SECONDARY OUTCOMES:
Patient survival | 5 years posttransplant
  patient survival 5 years posttransplant will be analyzed
Graft survival | 5 years posttransplant
  Graft survival 5 years posttransplant will be analyzed
Graft function and proteinuria | 5 years posttransplant
  5-year graft function will be analyzed by serum creatinine and measured creatinine clearance, proteinuria by proteinuria within a 24h urine collection period
Graft function | 5 years posttransplant
  5-year graft function will be analyzed by serum creatinine and measured creatinine clearance, proteinuria by proteinuria within a 24h urine collection period
Graft function | 5 years posttransplant
  5-year graft function will be analyzed by measured creatinine clearance
Proteinuria | 5 years posttransplant
  5-year proteinuria will be analyzed urine collected 24 hours
Incidence of acute rejection | 1 year posttransplant
  incidence of biopsy proven acute rejection within 1 year posttransplant will be analyzed
Incidence of acute rejection | 2 years posttransplant
  incidence of biopsy proven acute rejection within 2 years posttransplant will be analyzed
Incidence of acute rejection | 5 years posttransplant
  incidence of biopsy proven acute rejection within 5 years posttransplant will be analyzed
Incidence of chronic allograft dysfunction | 5 years posttransplant
  Chronic allograft dysfunction (progressive decline of graft function) will be analyzed at 5 years posttransplant.
Incidence of severe infectious disease | 5 years posttransplant
  severe infectious disease as defined by need for in-hospital treatment
Incidence of malignancy | 5 years posttransplant
  all types of malignancies within 5 years posttransplant will be evaluated
Incidence of side effects associated with Rtx | 5 years posttransplant
  all side effects of Rtx treatment which have been described in literature, will be listed

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Weimer, Prof. Dr., Principal Investigator — University of Giessen, Department of Internal Medicine
Locations (1):
- Department of Internal Medicine, University of Giessen, Giessen, Germany

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data are available to the members of the study group who treat the patients in the Department of Internal Medicine, University Clinic of Giessen (i.e. all participants of the study group working in the Department of Internal Medicine)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data will be available up to 1year post study completion
Access Criteria: seen above

REFERENCES:
- [Background] Hackstein H, Renner FC, Bohnert A, Nockher A, Frommer T, Bein G, Weimer R. Dendritic cell deficiency in the blood of kidney transplant patients on long-term immunosuppression: results of a prospective matched-cohort study. Am J Transplant. 2005 Dec;5(12):2945-53. doi: 10.1111/j.1600-6143.2005.01101.x. PMID 16303009
- [Background] Sadeghi M, Daniel V, Weimer R, Wiesel M, Hergesell O, Opelz G. Differential early posttransplant cytokine responses in living and cadaver donor renal allografts. Transplantation. 2003 Apr 27;75(8):1351-5. doi: 10.1097/01.TP.0000063706.52369.ED. PMID 12717229
- [Background] Staak A, Renner F, Suesal C, Dietrich H, Rainer L, Kamali-Ernst S, Ernst W, Padberg W, Opelz G, Weimer R. Immunoglobulin induction therapy in renal transplant recipients: Effects on immunoglobulin and regulatory antibody levels. Transplant Proc. 2006 Dec;38(10):3483-5. doi: 10.1016/j.transproceed.2006.10.041. PMID 17175311
- [Background] Weimer R, Melk A, Daniel V, Friemann S, Padberg W, Opelz G. Switch from cyclosporine A to tacrolimus in renal transplant recipients: impact on Th1, Th2, and monokine responses. Hum Immunol. 2000 Sep;61(9):884-97. doi: 10.1016/s0198-8859(00)00152-x. PMID 11053632
- [Background] Weimer R, Mytilineos J, Feustel A, Preiss A, Daniel V, Grimm H, Wiesel M, Opelz G. Mycophenolate mofetil-based immunosuppression and cytokine genotypes: effects on monokine secretion and antigen presentation in long-term renal transplant recipients. Transplantation. 2003 Jun 27;75(12):2090-9. doi: 10.1097/01.TP.0000058808.37349.23. PMID 12829918
- [Background] Weimer R, Staak A, Susal C, Streller S, Yildiz S, Pelzl S, Renner F, Dietrich H, Daniel V, Rainer L, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. ATG induction therapy: long-term effects on Th1 but not on Th2 responses. Transpl Int. 2005 Feb;18(2):226-36. doi: 10.1111/j.1432-2277.2004.00047.x. PMID 15691277
- [Background] Weimer R, Susal C, Yildiz S, Staak A, Pelzl S, Renner F, Dietrich H, Daniel V, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. Post-transplant sCD30 and neopterin as predictors of chronic allograft nephropathy: impact of different immunosuppressive regimens. Am J Transplant. 2006 Aug;6(8):1865-74. doi: 10.1111/j.1600-6143.2006.01407.x. Epub 2006 Jun 9. PMID 16771810
- [Background] Daniel V, Naujokat C, Sadeghi M, Renner FC, Weimer R, Opelz G. Association of high IFN-gamma plasma levels with low B-cell counts in renal transplant recipients with stable long-term graft function. Clin Transplant. 2010 Mar-Apr;24(2):281-9. doi: 10.1111/j.1399-0012.2009.01067.x. Epub 2009 Aug 27. PMID 19712086
- [Background] Susal C, Dohler B, Opelz G. Graft-protective role of high pretransplantation IgA-anti-Fab autoantibodies: confirmatory evidence obtained in more than 4000 kidney transplants. The Collaborative Transplant Study. Transplantation. 2000 Apr 15;69(7):1337-40. doi: 10.1097/00007890-200004150-00021. PMID 10798750
- [Background] Susal C, Pelzl S, Dohler B, Opelz G. Identification of highly responsive kidney transplant recipients using pretransplant soluble CD30. J Am Soc Nephrol. 2002 Jun;13(6):1650-6. doi: 10.1097/01.asn.0000014256.75920.5b. PMID 12039995
- [Derived] Weimer R, Karakizlis H, Renner F, Dietrich H, Daniel V, Susal C, Schuttler C, Kamper D, Leicht D, Worlen M, Milchsack K, Renner L, Stich M, Grone HJ, Hecker A, Horbelt R, Padberg W, Opelz G. Long-term compromised immune regulation after rituximab induction in blood group incompatible (ABOi) living-donor renal transplantation - 5 year results of a prospective pilot study. Front Immunol. 2025 Dec 12;16:1706158. doi: 10.3389/fimmu.2025.1706158. eCollection 2025. PMID 41459482